CLINICAL TRIAL: NCT04408027
Title: Mental Health Support for SickKids Children and Families During COVID-19 Using Established eHealth Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Suneeta Monga, Associate Psychiatrist-In-Chief, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB1000070362
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Anxiety Disorder of Childhood or Adolescence
Keywords: anxiety disorder; child; adolescent; virtual-care; cognitive behavioural therapy; COVID-19; mental health
MeSH Terms: conditions — Anxiety Disorders; COVID-19; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The current study will leverage an adapted virtual-care cognitive behavioural therapy program for children with anxiety (VC-CBT). The VC-CBT protocol will involve 12 sessions (of one hour in duration) delivered by a CBT therapist using PHIPA (Personal Health Information Protection Act) compliant Zoom. An initial session will review therapy goals and psychoeducation about anxiety. Sessions 2 and 3 will focus on feeling identification and will introduce relaxation strategies. Sessions 4 and 5 will introduce cognitive distortions and restructuring strategies. Sessions 6 and 7 will introduce exposure tasks. Sessions 8 to 11 will involve practicing cognitive restructuring skills and completing exposures. The final session will review relapse prevention. Parents will participate in the first and last sessions, as well as join at the end of each session for a brief review of the skills learned during the session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual-Care Cognitive Behavioural Therapy (Experimental)
  Interventions: Behavioral: Virtual-Care Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Virtual-Care Cognitive Behavioural Therapy — The feasibility, participation barriers, and acceptability of the intervention, virtual-care cognitive behavioural therapy (VC-CBT), will be evaluated for children with anxiety. The VC-CBT protocol will involve 12 sessions (of one hour in duration) delivered by a CBT therapist using PHIPA (Personal Health Information Protection Act) compliant Zoom. An initial session will review therapy goals and psychoeducation about anxiety. Sessions 2 and 3 will focus on feeling identification and will introduce relaxation strategies. Sessions 4 and 5 will introduce cognitive distortions and restructuring strategies. Sessions 6 and 7 will introduce exposure tasks. Sessions 8 to 11 will involve practicing cognitive restructuring skills and completing exposures. The final session will review relapse prevention. Parents will participate in the first and last sessions, as well as join at the end of each session for a brief review of the skills learned during the session.

SUMMARY:
Coronavirus disease 2019 (COVID-19) and associated emergency measures (EM) have dramatically impacted the lives of children/adolescents (children) and families. The closure of schools, social and recreational activities, and modifications to work environments has led to significant changes in the way children and families are working, living and socializing. Although the impact on the mental health of children and families has not been well researched, it is anticipated that already stressed children and families with pre-COVID-19 mental health challenges are at significant risk for deterioration in their mental health. As such, the implementation, and evaluation (specifically: feasibility, acceptability and barriers) of virtual-care interventions to alleviate child and family anxiety and enhance family functioning are critical. Virtual-care also optimizes health equity initiatives in reducing social, economic and environmental barriers to services that can improve or maintain mental health (WHO, 2017; MOHLTC, 2018).

The current study will evaluate an adapted virtual-care cognitive behavioural therapy (CBT) program for children with anxiety (VC-CBT). CBT has a strong evidence-base in treating children with anxiety disorders (Higa-McMillan, Francis, Rith-Najarian, and Chorpita, 2016; Seligman and Ollendick, 2011), with increasing evidence supporting the efficacy of virtual-care CBT for childhood anxiety disorders (Carpenter, Pincus, Furr, and Comer, 2018; Slone, Reese, and McClellan, 2012). This study aims to evaluate the feasibility, participation barriers related to social determinants of health (SDH) and acceptability of this virtual-care intervention in addressing mental health challenges associated with the COVID-19 pandemic and ensuing EM in the immediate time-period. Early evaluation of this virtual-care intervention will enable future scale-up of this intervention during the post-pandemic recovery time-period and during subsequent COVID-19 waves, if necessary.

DETAILED DESCRIPTION:
Study Design: This is a pragmatic prospective pre-post feasibility study to assess whether virtual-care delivery of mental health interventions are acceptable and feasible with regard to recruitment and retention, participation barriers (inclusive of SDH barriers), child and parent acceptability, and adherence. Targeted symptoms of the intervention (e.g., child anxiety) will be evaluated as secondary outcomes to gather preliminary data on efficacy.

Estimated Sample Size: In this first feasibility phase, participants will include children referred for treatment to Psychiatry. For the purpose of this pragmatic trial, we aim to recruit 20 participants for this intervention. According to Hertzog, a sample size of 20 participants is adequate for pilot studies to examine intervention feasibility and to develop estimates of variance to compute power for larger studies (Hertzog, 2008).

Data Analyses: Data for demographic variables will be summarized using counts, percentages, measures of central tendency (mean, median, and mode) and measures of sample variation (standard deviation, range). Parametric statistics (mean, standard deviation) will be used for interval and ratio data. To assess the feasibility and acceptability of this intervention, results will include analyses of recruitment, social determinant barriers and adherence rates and responses to satisfaction/evaluation and alliance scales. Pre-post analysis will also include comparing mean changes in COVID specific distress, and intervention specific comparisons of child anxiety.

Knowledge Translation: Our integrated Knowledge-to-action (iKTA) approach has involved family, clinician and scientist engagement from the outset and will continue to do so. Participants will receive updates through e-newsletters and information through email. Knowledge gained will be presented at conferences and publications to further the impact of generating future hypothesis-driven research and funding support.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to 17 years old
* Meet criteria for anxiety disorder as primary diagnosis
* Parent(s)/primary caregiver(s) and children both proficient in English

Exclusion Criteria:

* Diagnosis of developmental delay
* Severity of comorbid psychopathology (e.g., bipolar disorder, psychosis) prohibits CBT as first-line treatment
* Lack of fluency in English (for parent(s)/primary caregiver(s) and/or children)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Participation Barriers | The Social Determinants of Health Questionnaire will be administered at baseline only, for each participant (approximately one week prior to the first of twelve sessions in the intervention).
  Participation barriers related to Social Determinants of Health (SDH) will be captured to assess intervention feasibility. Participation barriers will be captured using the Social Determinants of Health Questionnaire (unpublished).
Number of Eligible Participants | The number of participants that were eligible for the study will be captured through study completion, estimated at approximately 1 year.
  Number of participants that were eligible for the study.
Number of Participants Approached | The number of participants that were approached for the study will be captured through study completion, estimated at approximately 1 year.
  Number of participants that were approached for the study.
Number of Participants Consented | The number of participants that were consented for the study will be captured through study completion, estimated at approximately 1 year.
  Number of participants consented for the study.
Rates of Refusal | The rates of refusal for participation in the study will be assessed through study completion, estimated at approximately 1 year.
  Rates of refusal for participation in the study.
Reasons for Refusal | The reasons of refusal for participation in the study will be assessed through study completion, estimated at approximately 1 year.
  Reasons for refusal for participation in the study.
Number of Sessions Completed in Total | The average number of sessions completed in total, for each participant, will be assessed through study completion, estimated at approximately 1 year.
  The average number of sessions completed in total will be captured to evaluate intervention adherence.
Adherence Index | The adherence index, for each participant, will be assessed through study completion, estimated at approximately 1 year.
  The adherence index (calculated using the formula: sessions completed/total sessions scheduled [sum of sessions attended, rescheduled, no-showed and cancelled]) will be used to evaluate intervention adherence.
Amount of time (in weeks) to complete the intervention | The amount of time (in weeks) to complete the intervention, for each participant, will be assessed through study completion, estimated at approximately 1 year.
  The amount of time (in weeks) to complete the intervention will be captured to evaluate intervention implementation experience.
Intervention Acceptability | The Virtual Care Satisfaction Survey will be administered once, within approximately one week after completion of the twelfth (final) intervention session (estimated to occur approximately 12 to 16 weeks after initiation of the study).
  The measure that will be used to assess the primary outcome of intervention acceptability is the Virtual Care Satisfaction Survey (Romanchych, unpublished).
Participant Satisfaction | The Virtual Care Satisfaction Survey will be administered once, within approximately one week after completion of the twelfth (final) intervention session (estimated to occur approximately 12 to 16 weeks after initiation of the study).
  The measure that will be used to assess participant satisfaction is the Virtual Care Satisfaction Survey (Romanchych, unpublished).
Working Alliance Inventory after First Intervention Session | The Working Alliance Inventory will be administered within approximately one week after completion of the first intervention session (estimated to occur approximately 1 to 2 weeks after initiation of the study).
  The Working Alliance Inventory will be used to assess participant satisfaction (WAI; Tracy & Kokotovic, 1989).
Working Alliance Inventory after Sixth Intervention Session | The Working Alliance Inventory will be administered within approximately one week after completion of the sixth intervention session (estimated to occur approximately 6 to 8 weeks after initiation of the study).
  The Working Alliance Inventory will be used to assess participant satisfaction (WAI; Tracy & Kokotovic, 1989).
Working Alliance Inventory after Final Intervention Session | The Working Alliance Inventory will be administered within approximately one week after completion of the twelfth (final) intervention session (estimated to occur approximately 12 to 16 weeks after initiation of the study).
  The Working Alliance Inventory will be used to assess participant satisfaction (WAI; Tracy & Kokotovic, 1989).

SECONDARY OUTCOMES:
Family Impact During a Pandemic at Baseline | CRISIS (parent/caregiver and youth forms) will be completed virtually by children and parents at baseline (approximately one week prior to the first of twelve sessions in the intervention).
  Coronavirus disease 2019 (COVID-19) specific distress will be assessed using the CoRonavIruS Health Impact Survey (CRISIS; Merikangas et al., unpublished) V0.1 Parent/Caregiver or Youth Baseline Form. Many items from this scale address social determinants of health, which will allow for understanding of family social determinants of health at baseline and over the course of the virtual-care treatment.
Family Impact During a Pandemic after Final Intervention Session | CRISIS forms will be completed virtually by children and parents, within approximately one week of completion of the twelfth (final) intervention session (approximately 12 to 16 weeks after initiation of the study).
  Coronavirus disease 2019 (COVID-19) specific distress will be assessed using the CoRonavIruS Health Impact Survey (CRISIS; Merikangas et al., unpublished) V0.1 Parent/Caregiver or Youth Follow-Up Form. Many items from this scale address social determinants of health, which will allow for understanding of family social determinants of health at baseline and over the course of the virtual-care treatment.
Efficacy of Virtual-Care CBT Intervention | The SCARED questionnaire will be completed at both baseline and within approximately one week after completion of the twelfth (final) intervention session (estimated to occur approximately 12 to 16 weeks after study initiation).
  To evaluate the efficacy of the virtual-care CBT intervention, change in child anxiety will be measured using child and parent-report Screen for Child Anxiety Related Disorders (SCARED; Birmaher et al., 1997). The SCARED is a child and parent self-report instrument used to screen for childhood anxiety disorders including general anxiety disorder, separation anxiety disorder, panic disorder and social phobia. In addition, it assesses symptoms related to school phobia. A total score of 25 of higher on the SCARED measure may indicate the presence of an anxiety disorder. Scores higher than 30 are more specific.
Clinician Virtual Care Experience | The Clinician Virtual Care Survey will be completed virtually by clinicians at both SickKids and CCMH at baseline.
  In order to evaluate the experience of clinicians (at The Hospital for Sick Children (SickKids) and the Centre for Community Mental Health (CCMH)) using virtual-care platforms during the work from home shift due to COVID-19 and to identify any challenges they may be facing, a Clinician Virtual Care Experience Survey (Romanchych, unpublished) will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Suneeta Monga, MD, FRCPC, Principal Investigator — The Hospital for Sick Children (SickKids)
Locations (1):
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Health Equity. Geneva; 2017.
- [Background] Ontario Ministry of Health and Long Term Care. Health Equity Guideline. Toronto, ON; 2018.
- [Background] Higa-McMillan CK, Francis SE, Rith-Najarian L, Chorpita BF. Evidence Base Update: 50 Years of Research on Treatment for Child and Adolescent Anxiety. J Clin Child Adolesc Psychol. 2016;45(2):91-113. doi: 10.1080/15374416.2015.1046177. Epub 2015 Jun 18. PMID 26087438
- [Background] Seligman LD, Ollendick TH. Cognitive-behavioral therapy for anxiety disorders in youth. Child Adolesc Psychiatr Clin N Am. 2011 Apr;20(2):217-38. doi: 10.1016/j.chc.2011.01.003. PMID 21440852
- [Background] Carpenter AL, Pincus DB, Furr JM, Comer JS. Working From Home: An Initial Pilot Examination of Videoconferencing-Based Cognitive Behavioral Therapy for Anxious Youth Delivered to the Home Setting. Behav Ther. 2018 Nov;49(6):917-930. doi: 10.1016/j.beth.2018.01.007. Epub 2018 Mar 5. PMID 30316490
- [Background] Slone NC, Reese RJ, McClellan MJ. Telepsychology outcome research with children and adolescents: a review of the literature. Psychol Serv. 2012 Aug;9(3):272-292. doi: 10.1037/a0027607. PMID 22867120
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Tracey T, Kokotovic A. Factor structure of the Working Alliance Inventory. Psychological Assessmen. Psychol Assess. 1989;1(3):207-210. doi:10.1037/1040-3590.1.3.207
- [Background] Birmaher B, Khetarpal S, Brent D, Cully M, Balach L, Kaufman J, Neer SM. The Screen for Child Anxiety Related Emotional Disorders (SCARED): scale construction and psychometric characteristics. J Am Acad Child Adolesc Psychiatry. 1997 Apr;36(4):545-53. doi: 10.1097/00004583-199704000-00018. PMID 9100430